CLINICAL TRIAL: NCT04618939
Title: Double Blind, Randomized Phase III Study to Evaluate the Immunogenicity and Safety of 'BR-TD-1001' Administered Intramuscularly in Healthy Children
Brief Title: To Evaluate the Immunogenicity and Safety of 'BR-TD-1001' Administered Intramuscularly in Healthy Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BR-TD-1001-CH-301
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Diphtheria; Tetanus
Keywords: Diphtheria; Tetanus
MeSH Terms: conditions — Diphtheria; Tetanus

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BR-TD-1001 (Experimental): Randomized subjects were assigned to receive a single dose of BR-TD-1001
  Interventions: Biological: BR-TD-1001
- Td-pur inj (Active Comparator): Randomized subjects were assigned to receive a single dose of Td-pur inj
  Interventions: Biological: Td-pur inj

INTERVENTIONS:
Biological: BR-TD-1001 — 0.5 mL, IM
  Arms: BR-TD-1001
Biological: Td-pur inj — 0.5 mL, IM
  Arms: Td-pur inj

SUMMARY:
The purpose of this study is to evaluate immunogenicity by measuring the seroprotection rate against diphtheria and tetanus at 28 days after vaccination with BR-TD-1001 and Td-pur-inj.

DETAILED DESCRIPTION:
Primary objective:

To evaluate immunogenicity by measuring the seroprotection rate against diphtheria and tetanus at 28 days after vaccination with BR-TD-1001 and Td-pur-inj.

Secondary objectives:

* To evaluate immunogenicity by measuring the geometric mean titer (of diphtheria and tetanus antitoxins at 28 days after vaccination with BR-TD-1001 and Td-pur-inj.
* To evaluate a boosting response by comparing before and after the administration through measurement of diphtheria and tetanus antitoxin titers at 28 days after vaccination with BR-TD-1001 and Td-pur-inj.
* To evaluate safety by observing solicited local and systemic adverse events that have occurred for 7 days after vaccination with BR-TD-1001 and Td-pur-inj.
* To evaluate safety by observing unsolicited adverse events that have occurred for 28 days after vaccination with BR-TD-1001 and Td-pur-inj.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy boys and girls aged 10 to 12 years
2. Those who received primary immunization (5 doses of diphtheria and tetanus vaccination until the age of 6)
3. Voluntary written consent of the subject and the legally acceptable representative(LAR) to participate in this clinical study

Exclusion Criteria:

1. 2 weeks have not passed since recovery from an acute disease
2. Temporary thrombocytopenia or neurological complications due to diphtheria or tetanus vaccination
3. History of a severe allergy to any component of the investigational product
4. History of a severe adverse event due to administration of diphtheria, tetanus, or diphtheria tetanus combined vaccine
5. Administration of tetanus, diphtheria, or diphtheria tetanus combined vaccine within 5 years
6. Unable to verify diphtheria and tetanus vaccination completed until the age of 6
7. History of infection with diphtheria or tetanus (if clinically, serologically or microbiologically confirmed)
8. Current chronic disease that impedes implementation or completion of the clinical study
9. Scheduled surgery during the study period
10. Acute fever with a tympanic temperature exceeding 38.0ºC within 72 hours before administration of the investigational vaccine
11. Administration of other vaccines within 28 days before screening
12. Use of immunosuppressants or immune modifying drugs within 3 months before screening
13. Those who have received immunoglobulin therapies or blood derived products within 3 months before screening, or are expected to receive them during the study period
14. Use of antipyretics/analgesics/nonsteroidal anti inflammatory drugs within 4 hours before administration of the investigational vaccine
15. Participation in other clinical studies within 28 days before screening
16. Those who were determined by the investigator to be ineligible for other reasons

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 218 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
The seroprotection rate of anti-diphtheria toxoid (DT) and anti-tetanus toxoid (TT) at 28 days after vaccination with the investigational products | 28 days after vaccination
  Seroprotection was defined as anti-DT and anti-TT antibody concentrations ≥ 0.1 IU/mL (ELISA)

SECONDARY OUTCOMES:
The geometric mean titer (GMT) of anti-DT and anti-TT at 28 days after vaccination with the investigational products | 28 days after vaccination
The boosting response for antitoxins of diphtheria and tetanus at 28 days after vaccination with the investigational product | 28 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jong Hyun Kim, Study Chair — Saint Vincent's Hospital, Korea
Locations (9):
- South Korea (9):
  - Changwon Fatima Hospital, Changwon
  - The Catholic University of Korea Daejeon St. Mary's Hospital, Daejeon
  - The Catholic University of Korea Incheon St. Mary's Hospital, Incheon
  - Asan Medical Center, Seoul
  - Eulji University Eulji General Hospital, Seoul
  - Hanil General Hospital, Seoul
  - Korea Cancer Center Hospital, Seoul
  - The Catholic University of Korea St. Paul's Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju

REFERENCES:
- [Derived] Choi UY, Kim KH, Lee J, Eun BW, Kim HM, Lee KY, Kim DH, Ma SH, Lee J, Kim JH. Immunogenicity and Safety of a Newly Developed Tetanus-Diphtheria Toxoid (Td) in Healthy Korean Adolescents: a Multi-center, Randomized, Double-blind, Active-Controlled Phase 3 Trial. J Korean Med Sci. 2021 Dec 20;36(49):e313. doi: 10.3346/jkms.2021.36.e313. PMID 34931494